CLINICAL TRIAL: NCT03470675
Title: Postpartum Perineal Pain After Obstetric Anal Sphincter Injuries: A Randomized Clinical Trial
Brief Title: Postpartum Perineal Pain After Obstetric Anal Sphincter Injuries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Feyce M. Peralta, MD, MS, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU00206016
Record Dates: First submitted 2018-03-02; First posted 2018-03-20 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Pain; Postpartum Depression
MeSH Terms: conditions — Pain; Depression, Postpartum | interventions — Sodium Chloride; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Epidural saline + IV saline (Placebo Comparator): Sterile saline via the epidural catheter. Sterile saline via intravenous catheter.
  Interventions: Drug: Epidural saline + IV saline
- Epidural morphine 3 mg + IV saline (Active Comparator): 3 milligrams morphine via the epidural catheter. Sterile saline via intravenous catheter.
  Interventions: Drug: Epidural morphine 3 mg + IV saline
- Epidural morphine 3 mg + IV ketamine 0.3 mg/kg (Active Comparator): 3 milligrams morphine via the epidural catheter. Ketamine 0.3 milligrams per kilogram via intravenous catheter.
  Interventions: Drug: Epidural morphine 3 mg + IV ketamine 0.3 mg/kg

INTERVENTIONS:
Drug: Epidural saline + IV saline — Sterile saline injection in the epidural catheter and in the intravenous catheter
  Arms: Epidural saline + IV saline
Drug: Epidural morphine 3 mg + IV saline — Morphine 3 milligrams injection in the epidural catheter and sterile normal saline intravenous catheter
  Arms: Epidural morphine 3 mg + IV saline
Drug: Epidural morphine 3 mg + IV ketamine 0.3 mg/kg — Morphine 3 milligrams injection in the epidural catheter and 0.3 milligrams per kilogram weight infused in the intravenous catheter
  Arms: Epidural morphine 3 mg + IV ketamine 0.3 mg/kg

SUMMARY:
Obstetric anal sphincter injuries (OASIS) encompass both third and fourth degree perineal tears. These tears can have a significant impact on women's quality of life in the short and long term. One of the most distressing immediate complications of this severe perineal injury is perineal pain. Women can also experience postpartum depression, dyspareunia, and altered sexual function after OASIS.

This is a randomized controlled trial to study the effects of three interventions (placebo, low dose intravenous ketamine plus epidural morphine, or epidural morphine alone) on acute pain after OASIS.

The objective of this study is to assess the incidence of perineal pain in postpartum patients 1 week after obstetric anal sphincter injuries.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years of age
* English-speaking
* Vaginal delivery (spontaneous or assisted)
* A full-term fetus (>37 weeks' gestation)
* OASIS as assessed by obstetrical provider
* Functional epidural analgesia at time of delivery
* Patient amenable to follow-up in specialty perineal clinic within the first week postpartum

Exclusion Criteria:

* Previous pelvic surgery
* History of chronic pelvic pain
* History of recurrent urinary tract infections
* Women with known malformations of their urinary tract
* True allergies to ketamine and/or morphine
* Preeclampsia or hypertensive disorder at the time of delivery
* Obstructive sleep apnea

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Perineal pain in postpartum patients 1 week after obstetric anal sphincter injuries. | 1 week after vaginal delivery
  Perineal pain 1 week after vaginal delivery measured using the VRS (verbal rating scale). The scale is scored 0 no pain and 10 highest pain.

SECONDARY OUTCOMES:
Perineal Pain | Day 1 after delivery
  Perineal pain day 1 after delivery using the McGill Pain Questionnaire (MPQ). This is a 15 question survey describing pain on a scale. The scale is scored 0 no pain and 3 severe pain.Combined score 0 low and 45 high pain.
Perineal Pain | 1 week after delivery
  Perineal pain day 7 after delivery using the McGill Pain Questionnaire (MPQ). This is a 15 question survey describing pain on a scale. The scale is scored 0 no pain and 3 severe pain.Combined score 0 low and 45 high pain.
Perineal Pain | 6 weeks after delivery
  Perineal pain 6 weeks after delivery using the McGill Pain Questionnaire (MPQ). This is a 15 question survey describing pain on a scale. The scale is scored 0 no pain and 3 severe pain.Combined score 0 low and 45 high pain.
Perineal Pain | 3 months after delivery
  Perineal pain 3 months after delivery using the McGill Pain Questionnaire (MPQ). This is a 15 question survey describing pain on a scale. The scale is scored 0 no pain and 3 severe pain.Combined score 0 low and 45 high pain.
Perineal Pain | 6 months after delivery
  Perineal pain 6 months after vaginal delivery measured using the VRS (verbal rating scale). The scale is scored 0 no pain and 10 highest pain.
Perineal Pain | 1 year after delivery
  Perineal pain 1 year after vaginal delivery measured using the VRS (verbal rating scale). The scale is scored 0 no pain and 10 highest pain.
Presence of postpartum depression | 1 week after delivery
  Presence of postpartum depression 7 days after delivery determined by using the Edinburgh Postnatal Depression Scale questionnaire. The questionnaire uses 10 questions scored 0 low to 3 high for a total score of 0 low 30 high. High scores indicate potential for depression.
Presence of postpartum depression | 6 weeks after delivery
  Presence of postpartum depression 6 weeks after delivery determined by using the Edinburgh Postnatal Depression Scale questionnaire. The questionnaire uses 10 questions scored 0 low to 3 high for a total score of 0 low 30 high. High scores indicate potential for depression.
Assessment of maternal-infant bonding | 1 week after delivery
  Assessment of maternal infant bonding using the Maternal Postnatal Attachment Scale (MPAS) questionnaire. 19 total question survey which is scored 1= low attachment and 5 = high attachment for each question. Total scores 19 low attachment to 95 high maternal infant attachment.
Assessment of maternal-infant bonding | 6 weeks after delivery
  Assessment of maternal infant bonding using the Maternal Postnatal Attachment Scale (MPAS) questionnaire. 19 total question survey which is scored 1= low attachment and 5 = high attachment for each question. Total scores 19 low attachment to 95 high maternal infant attachment.
Assessment of maternal-infant bonding | 3 months after delivery
  Assessment of maternal infant bonding using the Maternal Postnatal Attachment Scale (MPAS) questionnaire. 19 total question survey which is scored 1= low attachment and 5 = high attachment for each question. Total scores 19 low attachment to 95 high maternal infant attachment.
Medoc Pathway Device Score | 1 week post delivery
  Medoc Pathway Device (Durham NC) pain sensory results using VRS (verbal rating scale) 0 = no pain and 10 = worst pain imaginable
Maternal quality of life | 3 months after delivery
  Patient Reported Outcome Measurement Information System (PROMIS) 29 questionnaire. 28 question survey
Female sexual function | 3 months after delivery
  Female Sexual Function Index questionnaire (FSFI).This is a 19 question survey which is scored 2 low sexual function and 36 high sexual function.
Promis 29 profile | 6 week
  29 question recovery survey, 28 questions scored 1 low to 5 high and one question scored 0-10 for pain. Low combined total score (poor) 28 High combine 150 total score (good)
Promis 29 profile | 3 month
  29 question recovery survey, 28 questions scored 1 low to 5 high and one question scored 0-10 for pain. Low combined total score (poor) 28 High combine 150 total score (good)
Brief Pain Inventory (Short Form) Modified | 1 day after delivery
  7 question survey. 6 items scored 0 no pain -10 worst pain you can imagine scale. 1 item scored as relief%. 0= no relief (poor) and 100% complete relief (good)
Brief Pain Inventory (Short Form) Modified | 1 week after delivery
  7 question survey. 6 items scored 0 no pain -10 worst pain you can imagine scale. 1 item scored as relief%. 0= no relief (poor) and 100% complete relief (good)
Brief Pain Inventory (Short Form) Modified | 6 weeks after delivery
  7 question survey. 6 items scored 0 no pain -10 worst pain you can imagine scale. 1 item scored as relief%. 0= no relief (poor) and 100% complete relief (good)
Brief Pain Inventory (Short Form) Modified | 3 months after delivery
  7 question survey. 6 items scored 0 no pain -10 worst pain you can imagine scale. 1 item scored as relief %. 0= no relief (poor) and 100% complete relief (good)

CONTACTS AND LOCATIONS:
Overall Officials: Feyce Peralta, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harvey MA, Pierce M, Alter JE, Chou Q, Diamond P, Epp A, Geoffrion R, Harvey MA, Larochelle A, Maslow K, Neustaedter G, Pascali D, Pierce M, Schulz J, Wilkie D, Sultan A, Thakar R; Society of Obstetricians and Gynaecologists of Canada. Obstetrical Anal Sphincter Injuries (OASIS): Prevention, Recognition, and Repair. J Obstet Gynaecol Can. 2015 Dec;37(12):1131-48. doi: 10.1016/s1701-2163(16)30081-0. PMID 26637088
- [Background] Macarthur AJ, Macarthur C. Incidence, severity, and determinants of perineal pain after vaginal delivery: a prospective cohort study. Am J Obstet Gynecol. 2004 Oct;191(4):1199-204. doi: 10.1016/j.ajog.2004.02.064. PMID 15507941
- [Background] Chang SR, Chen KH, Lee CN, Shyu MK, Lin MI, Lin WA. Relationships between perineal pain and postpartum depressive symptoms: A prospective cohort study. Int J Nurs Stud. 2016 Jul;59:68-78. doi: 10.1016/j.ijnurstu.2016.02.012. Epub 2016 Feb 26. PMID 27222452
- [Background] Bauchat JR, Higgins N, Wojciechowski KG, McCarthy RJ, Toledo P, Wong CA. Low-dose ketamine with multimodal postcesarean delivery analgesia: a randomized controlled trial. Int J Obstet Anesth. 2011 Jan;20(1):3-9. doi: 10.1016/j.ijoa.2010.10.002. PMID 21224020